CLINICAL TRIAL: NCT06418295
Title: Cytokine Alterations Associated With Persistent Post-surgical Pain and Their Regulation Through Epigenetic Changes - A Pilot Study
Brief Title: Cytokine Alterations and Chronic Post-Surgical Pain
Status: Not yet recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Abhijit Biswas, Anesthesiologist, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: CPSP Epigenetics
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Chronic Post Operative Pain
Keywords: chronic pain; epigentics
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (7 mL) collected at the following time points:
  1. Pre-operatively before surgery.
  2. Post-operative day 1 following surgery
  3. 3 months following surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Unilateral thoracotomy: Unilateral thoracotomy to proceed according to standard of care guidelines.
  Interventions: Other: Unilateral thoracotomy

INTERVENTIONS:
Other: Unilateral thoracotomy — Unilateral thoracotomy to proceed as per standard of care guidelines. Thoracic epidural analgesia, or patient controlled analgesia (PCA) pumps will be offered to each study participant as per standard of care. Pre- and post-operative (post-operative day 1 and 3 months) pain scores and blood samples will be collected. Blood samples will be analyzed to determine the concentration of cytokines, chemokines, and growth factors that are potentially associated with CPSP (epidermal growth factor, eotaxin, fibroblast growth factor basic, G-CSF, GM-CSF, human growth factor, IFN-α, IFN-γ, IL-1ra, IL-1β, IL-2, IL-2r, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12 (p40/p70), IL-13, IL-15, IL-17, IP-10, MCP-1, MIG, MIP-1α, MIP-1β, RANTES, TNF-α, and VEGF). DNA promotor methylation for these targets will also be investigated.

SUMMARY:
Chronic Post-Surgical Pain (CPSP) is a condition that involves experiencing pain and/or discomfort that lasts for more than 3 months following surgery without any explainable cause of this pain such chronic infection or pain caused from a condition preceding surgery. This condition negatively impacts health related quality of life and is associated with significant financial burden both for the patient and health care system. Patients undergoing common surgeries such as amputation, breast surgery, hernia repair, coronary artery bypass, and caesarean section can be prone to developing CPSP. CPSP may be caused by the release and expression of different cellular molecules called cytokines and chemokines that can cause a pain response when they are present in the body at certain levels. After surgical incision, tissue cells have been shown to release cytokines and chemokines, thus increasing the concentration of these molecules in the patient's blood. It is not entirely known what mechanisms cause the increased expression of chemokines and cytokines. One method that may play a role in in this expression is epigenetics which is the alteration of gene expression without permanently altering the structure of DNA. Unlike mutations, epigenetic changes are dynamic, possibly reversible, and are influenced by environmental and behavioral changes such as diet, exercise, disease, stress, toxin exposure etc. Epigenetic changes occur all throughout our life and have been associated with several disease processes such as cancer, diabetic complications, and chronic pain. At the molecular level, certain events take place that can regulate (increase or decrease) the expression of cytokines and chemokines, most notably DNA methylation of their promotor (which involves adding molecules to DNA that does not change its structure but changes it's activity). The investigators are conducting this study to determine if the alteration of specific cytokines are associated with the occurrence of CPSP and whether these cytokines are regulated by DNA methylation at their promoter. This study will take place at London Health Sciences Centre and will recruit up to 60 patients who will be undergoing a thoracotomy procedure (surgery of the chest area).

DETAILED DESCRIPTION:
Chronic Post-Surgical Pain (CPSP), defined by the International Association for the Study of Pain, is a clinical discomfort that lasts more than 3 months post-surgery without other causes of pain such as chronic infection or pain from a chronic condition preceding the surgery. This condition negatively impacts health related quality of life and is associated with significant financial burden both for the patient and health care system. Patients undergoing a multitude of procedures, from amputation to hernia repair, are prone to develop CPSP with variable incidences.

CPSP may be a result of peripheral and central sensitization triggered by the release of cytokines and chemokines following surgery due to possible alterations in genetic expression. At the cellular level, after surgical incision, tissue cells from local areas have been implicated to drive synthesis of such cytokines/chemokines leading to alterations of their serum levels, including nerve growth factors (NGF) and interleukins (IL-1β). Specific regulatory mechanisms leading to augmented synthesis of these cytokines in the context of CPSP remain elusive. Several regulatory mechanisms may influence production of each cytokine. One method is via epigenetic mechanisms, which are defined as the alteration of gene expression without any structural genomic alterations that may regulate cytokine production at the transcriptional and post transcriptional levels. Among these listed epigenetic mechanisms, DNA methylation has been well studied and plays a key role in translation4. In general, hypomethylation of the promoter region leads to increased gene expression and vice versa. In this study the investigators wish to investigate how these mechanisms could be implicated in the expression of cytokines and chemokines in CPSP.

Patients undergoing unilateral thoracotomy will be included in this study. Their surgery and follow up care will proceed according to standard of care guidelines. Thoracic epidural analgesia, or patient controlled analgesia (PCA) pumps will be offered to each study participant as per standard of care. Patients' pain will be assessed preoperatively and postoperatively on day 1 and 3 months. Blood samples will also be taken during these times points and analyzed to determined the concentrations of the following cytokines, chemokines and growth factors:epidermal growth factor, eotaxin, fibroblast growth factor basic, G-CSF, GM-CSF, human growth factor, IFN-α, IFN-γ, IL-1ra, IL-1β, IL-2, IL-2r, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12 (p40/p70), IL-13, IL-15, IL-17, IP-10, MCP-1, MIG, MIP-1α, MIP-1β, RANTES, TNF-α, and VEGF. The occurrence of DNA methylation at the promotor region of these targets will be assessed via polymerase chain reaction (PCR) analysis. Results of these postoperative analyses will be compared to pre-operative molecular concentrations and pain scores to determine the association between epigenetic modifications (if any) and the development of CPSP and whether these modifications are driven by DNA promotor methylation.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Undergoing unilateral thoracotomy for the first time on that side
3. Willing to provide informed consent for study participation.
4. Patient with malignancy that needs thoracotomy for surgical resection.

Exclusion Criteria:

1. Chronic pain prior to surgery
2. Pre-existing fibromyalgia
3. Long-term opioid use
4. Diabetes mellitus
5. Inflammatory bowel disease
6. Pre-existing neurological disease
7. Pre-existing nerve injury
8. Evidence of dementia, delirium or cognitive disorder that may interfere with study participation
9. Malignancy other than lung cancer
10. Autoimmune disorder (e.g. rheumatoid arthritis and psoriatic arthritis)
11. Pregnancy
12. Inability to communicate in the English language (required for completion of questionnaires and provision of pain scores).
13. Patents on antiepileptic medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled to undergo thoracotomy for malignancy at Victoria Hospital, London Health Science Centre.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of temporal alterations of cytokines in patients with CPSP. | 3 months
  Cellular assays will be performed on blood samples obtained pre-and postoperatively to determined the level of expression of certain chemokines, cytokines, and growth factors that have been shown to be potentially related to CPSP. Pre and postoperative results will be compared to determine the association that each may have on the development of CPSP.
Identification of specific DNA promoter methylation regulating production of specific cytokines | 3 months
  Cellular assays will be performed on blood samples obtained pre-and postoperatively to determine if DNA promotor methylation is associated with changes in expression of the cytokines being investigated. Pre and postoperative results will be compared to determine the impact that this potential epigenetic change (DNA promotor methylation) may have on the development of CPSP.
Generate initial data to determine the sample size needed to adequately power a larger trial | 3 months
  As this is a pilot study, data will be analyzed to determine the sample size needed to power a larger, randomized controlled trial.

CONTACTS AND LOCATIONS:
Overall Officials: Abhijit Biswas, Principal Investigator — Western University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macrae WA, Davies HTO, Crombie IK, Linton S, Croft P, Von Korff M, LeResche L. Chronic postsurgical pain, Epidemiology of Pain, 1999, Seattle International Association for the Study of Pain (pg. 125-42)
- [Background] Macrae WA. Chronic post-surgical pain: 10 years on. Br J Anaesth. 2008 Jul;101(1):77-86. doi: 10.1093/bja/aen099. Epub 2008 Apr 22. PMID 18434337
- [Background] Richebe P, Capdevila X, Rivat C. Persistent Postsurgical Pain: Pathophysiology and Preventative Pharmacologic Considerations. Anesthesiology. 2018 Sep;129(3):590-607. doi: 10.1097/ALN.0000000000002238. PMID 29738328
- [Background] Aroke EN, Joseph PV, Roy A, Overstreet DS, Tollefsbol TO, Vance DE, Goodin BR. Could epigenetics help explain racial disparities in chronic pain? J Pain Res. 2019 Feb 18;12:701-710. doi: 10.2147/JPR.S191848. eCollection 2019. PMID 30863142
- [Background] Descalzi G, Ikegami D, Ushijima T, Nestler EJ, Zachariou V, Narita M. Epigenetic mechanisms of chronic pain. Trends Neurosci. 2015 Apr;38(4):237-46. doi: 10.1016/j.tins.2015.02.001. Epub 2015 Mar 9. PMID 25765319
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820